CLINICAL TRIAL: NCT03274596
Title: Effect of Vitamin E Supplementation on Oxidative Stress and Retinopathy of Prematurity in Preterm Infants <1500 g: A Randomized Clinical Trial.
Brief Title: Effect of Vitamin E for Prevention of Retinopathy of Prematurity: A Randomized Clinical Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Perinatologia Isidro Espinosa de los Reyes (Other Government)
Responsible Party: Principal Investigator, Silvia Romero-Maldonado, Principal Investigator, Instituto Nacional de Perinatologia Isidro Espinosa de los Reyes
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 212250-10231
Record Dates: First submitted 2017-09-04; First posted 2017-09-07 (Actual); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Retinopathy of Prematurity
Keywords: Oxidative Damage; Vitamin E; Total Antioxidant Capacity; Retinopathy of Prematurity
MeSH Terms: conditions — Retinopathy of Prematurity | interventions — Vitamin E

STUDY DESIGN:
Intervention Model Description: participants were randomly assigned to one of two treatmenst (A and B) using a computarized random number generator sequence; this process was handled by the hospital pharmacy staff. Group A: received vitamin E 12.5 IU orally every 12 hours, from 72 h after birth until 28 days of age, Group B: received orally sterile water (placebo) orally every 12 hours, from 72 h after birth until 28 days of age,
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The placebo was made by a pharmacologist and was the only person who knows the treatment of A and B. The placebo was administered by nursing staff and had the same appearance and amount as vitamin E. Neither the parents of the participants nor the researchers involved in the care or analysis of the data knew the content of the treatment and B until the end of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment A (Active Comparator): Group A: received 12.5 IU of vitamin E orally every 12 hours, from 72 h of birth to 28 days old.
  Interventions: Drug: Vitamin E
- Treatment B (Placebo Comparator): Group B: received 12.5 IU of placebo orally every 12 hours, from 72 hours of birth to 28 days old.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin E
  Arms: Treatment A
Drug: Placebo
  Arms: Treatment B

SUMMARY:
The retinopathy of prematurity (ROP) is a public health problem, the main causes of ROP are prematurity, use of oxygen, malnutrition and oxidative stress. Vitamin E was used beforehand however its use was stopped because of its association with sepsis and enterocolitis caused by the excipient of vitamin E. The purpose of this study is to use vitamin E to prevent ROP, without the previously used excipients.

DETAILED DESCRIPTION:
Antioxidant defence mechanisms include cellular and extracellular enzymes. Vitamin E is the main fat-soluble vitamin responsible for the protection of cell membranes against peroxidation, thus, it protects polyunsaturated fatty acids from peroxidation which is a step in the pathogenesis of ROP.

Previous research on the roles of vitamin E, in the prevention of BPD and ROP was halted because of complications involving sepsis and necrotising enterocolitis. These complications were caused by the compositions of vitamin E oral presentations, which contain polyethylene glycol, propylene glycol, ethanol and, polysorbate 80. These substances, which are used as excipients, may generate adverse effects in premature newborns. These preparations were not used in this project to avoid the development of necrotising enterocolitis, and because these formulations are not commercially available in Mexico.

The infants were randomly assigned to one of two groups using a computerized random number generator sequence; this process was handled by the hospital pharmacy staff. The treated group, received vitamin E 12.5 IU orally every 12 hours, from 72 h after birth until 28 days of age, the first blood sample collected from the newborns before the intervention was considered the baseline, and subsequent samples were obtained at 15 and 28 days of age.

Control group: received orally sterile water (placebo)

ELIGIBILITY:
Inclusion Criteria:

* Newborn weight < 1500 g
* Diagnosed respiratory distress syndrome (RDS)
* Patients who required mechanical ventilation or CPAP

Exclusion Criteria:

* Congenital malformations
* Rh incompatibility
* Non-immune or immune hydrops fetalis
* Intraventricular haemorrhage III/IV grade

Ages: 3 Days to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2015-10-01 (Actual); Study Completion 2015-12-01 (Actual)

PRIMARY OUTCOMES:
Incidence of retinopathy of prematurity | For the first retinopathy diagnosis, ophthalmological evaluation was performed at 28 days of birth.
  Retinopathy of prematurity was classified according to the International Classification of Retinopathy of Prematurity revisited 2005.

SECONDARY OUTCOMES:
Incidence of bronchopulmonary dysplasia (BPD) | Incidence of BPD was measured in each participant at 28 days old.
  BPD diagnosis was established according to the National Institute of Child Health and Human Development (NICHD) Workshop summary.
Severity of bronchopulmonary dysplasia (BPD) | Severity of BPD was measured at corrected 36 weeks' gestational age.
  Severity was classified into one of three stages: mild, when the patient did not required oxygen; moderate, when the patient required 30% oxygen; and severe when the patient required >30% oxygen, had nasal continuous positive airway pressure (CPAP), or mechanical ventilation.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Romero-Maldonado, M.Sc., Principal Investigator — Instituto Nacional de Perinatología Isidro Espinosa de los Reyes

REFERENCES:
- [Derived] Romero-Maldonado S, Montoya-Estrada A, Reyes-Munoz E, Guzman-Grenfell AM, Torres-Ramos YD, Sanchez-Mendez MD, Tolentino-Dolores M, Salgado-Valladares MB, Belmont-Gomez A, Najera N, Ceballos G, Cardona-Perez JA, Hicks JJ, Mancilla-Ramirez J. Efficacy of water-based vitamin E solution versus placebo in the prevention of retinopathy of prematurity in very low birth weight infants: A randomized clinical trial. Medicine (Baltimore). 2021 Aug 6;100(31):e26765. doi: 10.1097/MD.0000000000026765. PMID 34397821